CLINICAL TRIAL: NCT05946668
Title: The VAginal Microbiome as a BiomaRker of VagInal Health in Women With BreaSt CancEr (ARISE)
Brief Title: Evaluation of Vaginal Microbiome as a Biomarker for the Improvement of Vaginal Health in Women With Breast Cancer, ARISE Study
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Arthur, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-22295; NCI-2023-03368 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-06-26; First posted 2023-07-14 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (vaginal sample, questionnaires, records): Participants undergo vaginal specimen self-collection via vaginal swab collection kit, complete questionnaires, and have medical records reviewed on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo vaginal specimen self-collection via vaginal swab collection kit
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Medical records reviewed
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study evaluates vaginal microbiome as a biomarker to improve vaginal and sexual health in women with breast cancer receiving endocrine therapy. Breast cancer is the most common cancer in United States women, aside from skin cancers. Endocrine therapy is standard treatment for 70% of invasive breast cancers, significantly affecting sexual health and often causing women to change their course of treatment or cease sexual activity. Changes in the vaginal microbiome, which is the collection of all microorganisms, such as bacteria, fungi, and viruses, that naturally live on and inside the body, are implicated in menopausal-related sexual health symptoms, but the vaginal microbiome (and associated immune responses) has not been explored as a biomarker for sexual health changes in hormone-related sexual health symptoms in breast cancer. A biomarker is a biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease. Ribonucleic acid (RNA)-sequencing is a cost-effective method to analyze both human and microbial transcripts. The RNA that is sequenced from a standard biological sample such as a swab is a snapshot of the expression of many different cells and can be used to simultaneously measure the quantities of microbes, the overall expression of the human host, and the quantities of immune cells. Information gathered from this study may help researchers establish the vaginal microbiome as a biomarker and therapeutic target to improve the vaginal and sexual health of women with breast cancer receiving endocrine therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether individuals who experience vaginal dryness have a distinct microbiome prior to treatment from those who do not in a sample of breast cancer survivors initiating endocrine therapy.

EXPLORATORY OBJECTIVE:

I. Explore potential mechanisms of microbiome-associated vaginal toxicity through correlation with host gene expression and deconvolved immune cell abundances.

OUTLINE: This is an observational study.

Participants undergo vaginal specimen self-collection via vaginal swab collection kit, complete questionnaires, and have medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 years and older
* Non-metastatic, estrogen and/or progesterone positive, human epidermal growth factor (HER) 2 negative breast cancer who will be receiving endocrine therapy, including tamoxifen, aromatase inhibitor, or ovarian suppression
* Endocrine positive women who have received chemotherapy (adriamycin and cytoxan + taxol; taxotere and cytoxan) will still be eligible but must have completed their treatment

Exclusion Criteria:

* Triple negative breast cancer patients
* Human epidermal growth factor (HER) 2 positive breast cancer patients
* Metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer receiving endocrine therapy at the Stephanie Spielman Comprehensive Breast Center (SSCBC) at the Ohio State University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation of Lactobacillus to Prevotella Ratio (LPR) with vaginal dryness | Through study completion, an average of 1 year
  The LPR will be calculated by aggregating the Lactobacillus genus counts and dividing by the aggregated Prevotella genus counts. The vaginal dryness (binary, Vaginal Assessment Scale score <= 2 versus > 2) will be related to the LPR (continuous) by logistic regression. Will use a two-sided Mann-Whitney-Wilcoxon test with Monte Carlo simulation. Descriptive statistics (frequencies, percentages, means, medians) and correlations will be used to describe sociodemographic factors, clinical factors, and patient reported outcomes. Parametric and nonparametric tests of difference will be used to compare variables.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K Arthur, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu